CLINICAL TRIAL: NCT01923948
Title: A Randomized Placebo-Controlled Study of Whether Pre-operative Pregabalin 150 mg Will Improve Pain Control in Patients With Hepatocellular Carcinoma Undergoing Partial Hepatectomy
Brief Title: Preoperative Pain Control in Liver Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EHBHKY2013-001-09
Record Dates: First submitted 2013-08-09; First posted 2013-08-16 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Pain, Postoperative; Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Hepatectomy; randomized controlled trials(RCTs); Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative; Carcinoma, Hepatocellular | interventions — Pregabalin; Sugars; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregabalin (Active Comparator): Single, 150 mg pre-operative oral dose of Pregabalin
  Interventions: Drug: Pregabalin
- Sugar Pill (Placebo Comparator): Single, placebo pre-operative dose
  Interventions: Drug: Placebo (for Pregabalin)

INTERVENTIONS:
Drug: Pregabalin — One 150 mg oral dose of Pregabalin given before surgery
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Placebo (for Pregabalin) — One oral dose of placebo given before surgery
  Other Names: Sugar pill manufactured to mimic Pregabalin 150 mg tablet
  Arms: Sugar Pill

SUMMARY:
Pregabalin 150mg or placebo are administered 1 hour preoperatively in patients undergoing partial hepatectomy. Postoperatively, patients receive morphine as rescue analgesic. Morphine consumption in the first 48 hours is documented. Postoperative pain is measured by the visual analogue scale (VAS) score.

DETAILED DESCRIPTION:
Methods: In this Randomized Controlled Trial, patients undergoing partial hepatectomy will be administered a single pre-operative dose of Pregabalin or a placebo. Primary endpoints are as follows:

* Post-operative analgesic requirements
* Post-operative VAS scale (rated 0-10)
* Complications
* Post-operative antiemetic requirement
* Length of stay

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing partial hepatectomy

Exclusion Criteria:

* contraindication against pregabalin
* creatinine > 2.0 mg/dl
* GGT >165, AST >105, ALT >135
* peptic Ulcus
* haemorrhagic diathesis
* angina pectoris, myocardial infarction
* stroke
* bronchial asthma
* opioid abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Postoperative Opioid Consumption | 48 hours

SECONDARY OUTCOMES:
Postoperative Pain Scores on the Visual Analog Scale | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: li ai jun, MD, Study Chair — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, China